CLINICAL TRIAL: NCT02492867
Title: A Pilot Study of Response-Driven Adaptive Radiation Therapy for Patients With Locally Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2015.035; HUM00098202 (Other: University of Michigan); P01CA059827 (NIH)
Record Dates: First submitted 2015-06-30; First posted 2015-07-09 (Estimated); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Positron-Emission Tomography; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Response-driven Adaptive RT (Experimental): Patients will receive treatment 5 days per week, in once daily fractions, for 30 treatments with dose per fraction individually adapted over the final 9 treatments. Patients may also receive concurrent chemotherapy with Carboplatin and Paclitaxel. Patients may receive consolidation chemotherapy (carboplatin and paclitaxel) or immunotherapy (durvalumab) at the discretion of the medical oncologist.
  Interventions: Radiation: Response-driven Adaptive Radiation Therapy; Drug: Carboplatin; Drug: Paclitaxel; Device: FDG-PET; Device: V/Q SPECT; Drug: Durvalumab

INTERVENTIONS:
Radiation: Response-driven Adaptive Radiation Therapy
Drug: Carboplatin — AUC 2 concurrent with RT; AUC 6 during consolidation. Given IV
Drug: Paclitaxel — 40 mg/m^2 IV concurrent with RT; 200 mg/m^2 during consolidation. Given IV
Device: FDG-PET
  Other Names: Positron Emission Tomography Scan
Device: V/Q SPECT
  Other Names: Single-photon Emission Computed Tomography Scan
Drug: Durvalumab — 10 mg/kg during consolidation. Given IV

SUMMARY:
Successful treatment of lung cancer with radiation therapy requires that the physicians determine exactly where the tumor is in the patient's body and seek to limit any unnecessary radiation to normal parts of the body. This study is designed to apply functional imaging, Fluorodeoxyglucose-Positron Emission Tomography (FDG-PET) ("a PET scan") and Ventilation/Perfusion Single Photon Emission Computerized Tomography (V/Q SPECT) ("a perfusion scan"), before treatment and then again during treatment to see if this scanning helps predict how well the treatment works and how well the lung functions during treatment. FDG-PET is a modern technology that uses small amounts of a radioactive glucose (FDG) to make images of the whole body and areas of active cancer. V/Q SPECT is an image mapping tool that helps assess how well the lungs are working. A Computerized Tomography (CT) will also be performed along with both of these procedures to help the researchers see clearly where the cancer or the healthy lung is located.

The researchers are also doing blood and urine tests in this study to look for markers to see if this helps them determine the patient's risk of developing side effects from radiation to the lungs. The researchers hope by using these types of tests that they can have more information to help decrease the amount of toxicity patients have from this type of treatment. The researchers hope that this study will help them in the future to design radiation treatment plans that provide the best treatment for each individual patient.

DETAILED DESCRIPTION:
This is a pilot study to improve local tumor control while maintaining the same rate of treatment toxicity by adapting therapy to the uninvolved lung and esophagus while continuing to adapt therapy to the tumor for patients with Stage II/III NSCLC.

Lung cancer is the leading cause of cancer death in the United States and worldwide. In 2012, there were 226,160 new cases and 160,340 deaths related to lung cancer in the United States. Approximately, 80-85% of lung cancers are NSCLC (Non-small Cell Lung Cancer), and 40% of these are locally advanced (stage II/III) at diagnosis. The current standard of care for these patients is "one size fits all" RT (Radiation Therapy) with concurrent chemotherapy in uniform regimens. Even after concurrent chemoradiation, however, the five year overall survival was still about 15%; almost one half of the patients failed locally. At the same time, intensification of both radiotherapy and concurrent chemotherapy may result in excessive toxicity or incomplete treatment. Therefore, it is critical to tailor the treatment to each individual's sensitivity in combination with functional imaging guided response-driven treatment and biomarker guided individualized dose prescription, thus taking into consideration both the tumor and toxicity profile.

Evidence suggests that high-dose radiation has the potential to improve local-regional control and overall survival in patients treated with fractionated therapy with concurrent chemotherapy.

However, it is challenging to deliver high dose RT in the majority of patients with locally advanced NSCLC without exceeding doses to organs at risk and causing significant side effects.

Investigators hypothesized that they could develop safer and more effective therapy by adapting treatment to the individual patient's response. With respect to the tumor, investigators hypothesized, that they could improve outcome by redistributing dose to the more aggressive regions of the tumor, assessed using mid-treatment FDG-PET (Positron Emission Tomography) scanning. With respect to uninvolved organs, investigators need methods of estimating tolerable radiation doses for the individual patient rather than the population average. Such a strategy requires assessing both global and regional normal lung function and the technology to deliver dose in a manner that minimizes damage to functional lung and esophagus.

During-RT FDG-PET/CT potentially can provide important benefits to individual patients by intensifying dose to more resistent tumor, allowing early changes to alternative, more efficacious treatment or by avoiding the unnecessary toxicity related to ineffective therapy.

Patients will also undergo a during treatment V/Q SPECT (Single-photon Emission Computed Tomography) scan, as an adaptive plan based on during-treatment SPECT may further optimize PART (Personalized Adaptive Radiotherapy) to avoid high dose radiation to the well-functioning regions, and would thus decrease RILT (Radiation Induced Lung Toxicity).

The combination of pre- and during V/Q SPECT can classify the lung into different functional regions, and a strategy to give differential priority to the regions has been developed to minimize lung damage.

Investigators plan to continue to collect data on serum biomarkers to further refine their biophysical model with the ultimate goal of individualizing radiation dose prescription.

By identifying high risk patients and adjusting OAR (Organs at Risk) dose limits to the threshold of tolerance, investigators anticipate a significant reduction in the incidence of toxicity from UMCC 2007.123 (NCT01190527) without compromised tumor control by applying the model to optimize radiation planning.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have FDG-avid and pathologically proven Stage IIA-IIIB non-small cell lung cancer.
* Patients must be considered unresectable or inoperable.
* Patients must be 18 years of age or older.
* Patients must have a Karnofsky performance (A measure general well-being and activities of daily life. Scores range between 0 and 100 where 100 represents normal and 0 represents death.) of score > or = to 70.
* Patients must have adequate organ and marrow function.
* Patient must be willing to use effective contraception if female with reproductive capability.
* Patients must be informed of the investigational nature of this study and given written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients with any component of small cell lung carcinoma
* Patients with evidence of a malignant pleural or pericardial effusion
* Prior radiotherapy to the thorax such that composite radiation would significantly overdose critical structures, either per estimation of the treating radiation oncologist or defined by failure to meet normal tissue tolerance constraints
* Patients cannot tolerate concurrent chemotherapy
* Pregnant women are excluded from this study because radiation has the potential for teratogenic or abortifacient effects.
* Prisoners are excluded for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Jolly, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - University of Michigan Cancer Center, Ann Arbor, Michigan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients were enrolled but were never treated, 5 patients started treatment but did not complete
Groups:
- Response-driven Adaptive RT: Patients received treatment 5 days per week, in once daily fractions, for 30 treatments with dose per fraction individually adapted over the final 9 treatments. Patients may have also received concurrent chemotherapy with Carboplatin and Paclitaxel. Patients may have received consolidation chemotherapy (carboplatin and paclitaxel) or immunotherapy (durvalumab) at the discretion of the medical oncologist.
  Response-driven Adaptive Radiation Therapy
  Carboplatin: AUC 2 concurrent with RT; AUC 6 during consolidation. Given IV
  Paclitaxel: 40 mg/m^2 IV concurrent with RT; 200 mg/m^2 during consolidation. Given IV
  FDG-PET
  V/Q SPECT
  Durvalumab: 10 mg/kg during consolidation. Given IV
Period: Overall Study
Arm/Group | Response-driven Adaptive RT
Started | 47
Completed | 42
Not Completed | 5
Not completed — Alternate therapy | 1
Not completed — Withdrawal by Subject | 2
Not completed — Disease progression after treatment started | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Response-driven Adaptive RT
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 28
Age, Continuous [Median (Full Range); unit: years] | 66.4 [50 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 43
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients for Whom Treatment is Feasible.
Description: To determine the feasibility of the proposed adaptive treatment strategy, we will look at the number of patients for whom treatment is feasible. Treatment is feasible if we are able to deliver the full treatment, using the image based spatial replanning and complete the cytokine assays in a short enough timeframe to adapt radiation dose.
Time Frame: 6 weeks (30 treatments, 5 days per week)
Measure: Count of Participants; unit: Participants
Arm/Group | Response-driven Adaptive RT
Number analyzed (Participants) | 47
Participants | 40

2. Primary Outcome: The Number of Patients That Experience Grade 2 or Greater Lung Toxicity
Description: Lung toxicity will be graded using CTCAE v4.0. These will include, but not be limited to: cough, dyspnea, pneumonitis, radiation pneumonitis, and radiographic or clinical pulmonary fibrosis.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Response-driven Adaptive RT
Number analyzed (Participants) | 47
Participants
  cough | 8
  pneumonitis | 1
  Dyspnea | 6
  radiation pneumonitis | 0
  Pulmonary fibrosis | 1

3. Primary Outcome: The Number of Patients That Experience Grade 2 or Greater Esophageal Toxicity
Description: Esophageal toxicities will be graded using CTCAE v4.0. These will include, but not be limited to esophagitis.
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Response-driven Adaptive RT
Number analyzed (Participants) | 47
Participants
  Esophageal hemorrhage | 1
  Esophageal Pain | 9
  Esophagitis | 7

4. Primary Outcome: Comparison of Delivered Dose to Dose That Would Have Been Administered Using the Criteria Described in Protocol UMCC 2007.123 (NCT01190527)
Description: Investigators will generate the treatment plan (and hence dose to PET avid region) each patient would have received if they had been treated on protocol UMCC 2007.123 (NCT01190527), which redistributed dose to the PET avid region but not through normal tissue. These dose values will then be compared to the doses actually given to assess for any mean differences.
Time Frame: 6 weeks (30 treatments, 5 days per week)
Population: 47 participants from this trial and 15 from the previous trial, UMCC 2007.123
Measure: Mean (Standard Deviation); unit: average total physical dose (Gy)
Arm/Group | Response-driven Adaptive RT
Number analyzed (Participants) | 62
average total physical dose (Gy)
  UMCC 2007.123 study: number analyzed (Participants) | 15
  UMCC 2007.123 study | 80.4 (6.01)
  UMCC 2015.035 Study: number analyzed (Participants) | 47
  UMCC 2015.035 Study | 67.7 (7.7)

5. Secondary Outcome: Time to Local Progression
Description: Defined as the time from start of treatment to time of local/regional progression on PET, summarized with the Kaplan-Meier method.
Time Frame: Up to 60 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Response-driven Adaptive RT
Number analyzed (Participants) | 47
percentage of patients
  Locoregional progression-free survival at 1 year | 69.2 [57 to 84.1]
  Locoregional progression-free survival at 2 years | 47.9 [35.1 to 65.3]

6. Secondary Outcome: Overall Survival Time
Description: Defined as the time from start of treatment to death.
Time Frame: Up to 60 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Response-driven Adaptive RT
Number analyzed (Participants) | 47
percentage of patients
  Overall survival at 1 year | 82.8 [72.6 to 94.4]
  Overall survival at 2 year | 62.3 [49.6 to 78.3]

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 36 months after the last dose of study treatment. Data was collected during a 6 year period.
Arm/Group | Response-driven Adaptive RT
All-Cause Mortality (participants affected / at risk) | 22/47
Serious Adverse Events (participants affected / at risk) | 13/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Response-driven Adaptive RT (N=47)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial Flutter (Cardiac disorders) | 2 (2)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Lung infection (Infections and infestations) | 4 (4)
malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
non-cardiac chest pain (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
stroke (Nervous system disorders) | 1 (1)
vascular disorders- other, specify (Vascular disorders) | 1 (1) — ischemia cerbrovascular
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Response-driven Adaptive RT (N=47)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
cholecystitis (Hepatobiliary disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 41 (81)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 25 (38)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 31 (61)
Esophageal Pain (Gastrointestinal disorders) | 38 (62)
Esophagitis (Gastrointestinal disorders) | 39 (73)
Fatigue (General disorders) | 45 (90)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Clinical fibrosis (General disorders) | 2 (3)
Rib fracture (General disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
pericarditis (Cardiac disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 (13)
Altered mental status (Psychiatric disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Radiation recall reaction (Injury, poisoning and procedural complications) | 1 (1)
superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 7 (7)
Upper respiratory infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT02492867/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT02492867/ICF_001.pdf